CLINICAL TRIAL: NCT06574373
Title: New Theranostic Biomarkers of Intraductal Mucinous Neoplasm (IPMN) Progression to Pancreatic Cancer for Patients' Outcome Improvement
Brief Title: Identification of New Theranostic Biomarkers of Pancreatic Tumor Progression
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); University of Messina (Other)
Responsible Party: Principal Investigator, Carbone Carmine, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 6797; PNRR-MCNT2-2023-12377229 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: IPMN, Pancreatic
Keywords: IPMN; Pancreatic cancer; precancerous lesions
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Pancreatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Radiomics imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with IPMN/pancreatic cancer diagnosis: Patients with indolent IPMN, invasive IPMN, and IPMN associated with pancreatic cancer, depending on their clinical course.
  Interventions: Other: Blood Collection Protocol for Patients with Indolent, Invasive, and Pancreatic Cancer-Associated IPMN Based on Clinical Course and Surgical Intervention

INTERVENTIONS:
Other: Blood Collection Protocol for Patients with Indolent, Invasive, and Pancreatic Cancer-Associated IPMN Based on Clinical Course and Surgical Intervention — Blood will be collected from patients with indolent IPMN, invasive IPMN, and IPMN associated with pancreatic cancer, depending on their clinical course. Patients with indolent IPMN will be monitored by the gastroenterology units of their respective institutions, which will inform the patient. Patients with invasive IPMN and/or associated with cancer will undergo surgical resection as part of their standard clinical care, and blood will be collected after informed consent is obtained by the surgical teams at each institution.

SUMMARY:
Intraductal papillary mucinous neoplasms (IPMN) are one of the main precursor lesions of pancreatic ductal adenocarcinoma (PDAC), a lethal disease predicted to become the second leading cause of cancer-related deaths in Western societies within a decade. The mechanisms underlying IPMN progression are poorly understood. The goal of IPMN management is to reduce the risk of patient death due to progression to PDAC through primary and secondary prevention (namely, early diagnosis and risk-reducing surgery). High-risk IPMNs (i.e., high-grade or main duct IPMNs, which account for 57-90% of cases) are referred for surgical resection, while low-risk IPMNs (6-46%) undergo periodic follow-up aimed at monitoring the acquisition of morphological features associated with malignancy over time. However, the clinical management of IPMN remains a significant challenge because the distinction between high and low-risk progression is based on imaging and histological criteria that are not unequivocally recognized and do not take into account the underlying biology of lesions that appear similar but are associated with different clinical behaviors. Consequently, patient risk stratification is often inaccurate, leading to suboptimal treatment. Approximately 1-11% of low-risk IPMN patients assigned to clinical follow-up have developed PDAC. Therefore, it is of paramount importance to improve the understanding of the biology and malignant potential of IPMN to improve prognosis and clinical management of affected patients and guide them toward personalized therapeutic approaches. The availability of markers capable of stratifying IPMN based on their risk of progression to PDAC could enhance the current malignancy criteria assessed in clinical settings by more accurately identifying patients who strongly need surgical resection.

**Study Objective** The aim of this study is to identify and validate biomarkers capable of distinguishing between low-risk and high-risk IPMN progression to PDAC. These biomarkers would help more accurately identify IPMN patients who could benefit from therapeutic intervention and/or surgical resection in the future. The study will include patients with IPMN followed at Fondazione Policlinico Gemelli IRCCS Roma, Fondazione G. Pascale IRCCS Naples, Azienda Ospedaliera Universitaria Integrata Verona, and Azienda Ospedaliera Universitaria Integrata Messina.

DETAILED DESCRIPTION:
**AIM1.**

1. **Identification** of genes and biological pathways associated with IPMN malignant transformation. The investigators aim to explore the molecular dynamics of tumor progression, focusing on cellular heterogeneity and phenotypic transitions.
2. **Characterization of the microenvironment** to understand its role in IPMN progression. The investigators will collect archival samples from 240 patients across four centers.
3. **Identification and validation in plasma** of selected patients of differentially expressed markers in indolent IPMN, invasive IPMN, and PDAC.

**AIM2.** The investigators will develop knowledge-based tools for diagnosing and treating IPMN and at-risk populations.

**AIM3.** The investigators will validate the role of key genes in IPMN carcinogenesis using in vitro study models.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of indolent IPMN under monitoring;
* Diagnosis of malignant IPMN or resectable pancreatic adenocarcinoma with associated IPMN (previously untreated); Written informed consent; Male and female patients aged 18 years or older;

Exclusion Criteria:

-Inability to provide written informed consent or to trace patients for the retrospective study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years old with Pancreatic IPMN. This cohort will consist of IPMN tissues collected via Formalin-Fixed Paraffin-Embedded from patients who have either developed or have never developed pancreatic cancer associated with IPMN.
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of IPMNs tumorigenic progression with a molecular profile | 2 years
  Identification of participants with malignant transformation and at least two-fold expression change of a specific molecular profile respect to indolent IPMN.
  All data will be collected and statistics will be done for the correlation between gene expression markers and malignant transformation.

SECONDARY OUTCOMES:
Validation of the prognostic molecular profile identified in the primary objective in both archived tissue and plasma samples | 2 years
  Retrospective analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Carbone, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Gemelli, Roma
  - IRCCS Fondazione Policlinico Universitario A. Gemelli, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agostini A, Piro G, Inzani F, Quero G, Esposito A, Caggiano A, Priori L, Larghi A, Alfieri S, Casolino R, Scaglione G, Tondolo V, Cammarota G, Ianiro G, Corbo V, Biankin AV, Tortora G, Carbone C. Identification of spatially-resolved markers of malignant transformation in Intraductal Papillary Mucinous Neoplasms. Nat Commun. 2024 Mar 29;15(1):2764. doi: 10.1038/s41467-024-46994-2. PMID 38553466
- [Result] Tanaka M, Fernandez-Del Castillo C, Kamisawa T, Jang JY, Levy P, Ohtsuka T, Salvia R, Shimizu Y, Tada M, Wolfgang CL. Revisions of international consensus Fukuoka guidelines for the management of IPMN of the pancreas. Pancreatology. 2017 Sep-Oct;17(5):738-753. doi: 10.1016/j.pan.2017.07.007. Epub 2017 Jul 13. PMID 28735806
- [Result] Levink I, Bruno MJ, Cahen DL. Management of Intraductal Papillary Mucinous Neoplasms: Controversies in Guidelines and Future Perspectives. Curr Treat Options Gastroenterol. 2018 Sep;16(3):316-332. doi: 10.1007/s11938-018-0190-2. PMID 30196428
- [Result] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766